CLINICAL TRIAL: NCT00530621
Title: A Phase 2 Double-Blind Randomized Study of Oral Enzastaurin HCl Versus Placebo Concurrently With Pemetrexed (Alimta®) as Second-Line Therapy in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Enzastaurin Versus Placebo With Pemetrexed for Participants With Advanced or Metastatic Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9820; H6Q-MC-JCBT (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — enzastaurin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemetrexed + Enzastaurin (Experimental)
  Interventions: Drug: enzastaurin; Drug: pemetrexed
- Pemetrexed + Placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: pemetrexed

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) loading dose then 500 mg, oral, daily Cycle 1 (28 days), subsequent cycles 21 days, until disease progression
  Other Names: LY317615
  Arms: Pemetrexed + Enzastaurin
Drug: placebo — oral, daily
  Arms: Pemetrexed + Placebo
Drug: pemetrexed — 500 milligrams per square meter (mg/m^2), intravenous (IV), day 8 Cycle 1 (28 days), day 1 subsequent cycles (21 days), until disease progression
  Other Names: LY231514; Alimta

SUMMARY:
The purpose of this study is to determine if the combination of enzastaurin and pemetrexed can extend survival time without progression of disease for participants who have advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed diagnosis of NSCLC with locally advanced or metastatic disease which cannot be cured.
* Participants must have disease which progressed after 1 prior systemic cytotoxic chemotherapy regimen for advanced disease.
* At least 1 measurable lesion.
* Must have stopped all previous systemic therapies for cancer for at least 2 weeks prior to enrollment.
* Must be able to follow study guidelines and be able to show up for appointments.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Previous treatment with enzastaurin or pemetrexed.
* Concurrent administration of any other antitumor therapy.
* Inability to swallow tablets.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (25):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scarborough, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richardson, Texas
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gauting
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aviano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presented in the participant flow are the reasons participants discontinued from study treatment.
Groups:
- Pemetrexed + Enzastaurin: Enzastaurin 1125 milligrams (mg) loading dose [total 9 tablets (three 125-mg tablets administered orally 3 times a day)] on Day 1 followed by total dose of 500 mg enzastaurin (two 125-mg tablets administered orally 2 times a day) on Days 2 to 28, and pemetrexed 500 milligrams per square meter (mg/m^2) intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by total dose of 500 mg enzastaurin (two 125-mg tablets administered orally 2 times a day) on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Pemetrexed + Placebo: Placebo loading dose [total 9 tablets (3 tablets administered orally 3 times a day)] on Day 1 followed by 4 placebo tablets (2 tablets 2 times a day) on Days 2 to 28, and pemetrexed 500 mg/m^2 intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by 4 placebo tablets (2 tablets 2 times a day) on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Started | 80 | 80
Received at Least 1 Dose of Study Drug | 79 | 80
Completed | 0 | 0
Not Completed | 80 | 80
Not completed — Adverse Event | 11 | 8
Not completed — Physician Decision | 2 | 4
Not completed — Progressive Disease (PD) | 47 | 40
Not completed — Sponsor Decision | 12 | 15
Not completed — Subject Decision | 4 | 7
Not completed — Death | 3 | 6
Not completed — Not Treated Due to PD Prior to Dosing | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.21) | 61.6 (9.57) | 61.4 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 54 | 54 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 1 | 4
  White | 69 | 73 | 142
  East Asian | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  France | 19 | 19 | 38
  United States | 17 | 17 | 34
  Portugal | 5 | 11 | 16
  Germany | 21 | 19 | 40
  Italy | 11 | 9 | 20
  South Korea | 7 | 5 | 12
Disease Stage at Study Entry [Count of Participants; unit: Participants] — Disease stage describes how big the tumor is and how far it has spread from the site of origin. Stages ranged from Stage I to Stage IV. Stage III is further separated into Stage IIIA (cancer is locally advanced and spread to nearby lymph node) and Stage IIIB (cancer has spread to distant lymph nodes and invaded other organs like heart or esophagus). Stage IV has cancer spread throughout the body.
  Participants
    Stage IIIA | 3 | 3 | 6
    Stage IIIB | 16 | 23 | 39
    Stage IV | 61 | 54 | 115

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the first documented observation of disease progression or death from any cause. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive disease (PD) was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. PFS was censored at the date of the last objective progression-free disease assessment for participants who did not experience PD or death at the data inclusion cut-off date.
Time Frame: Baseline to measured progressive disease up to 9.92 months
Population: All randomized participants. Twenty five (25) participants in Pemetrexed + Enzastaurin group and twenty three (23) participants in Pemetrexed + Placebo group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 80 | 80
months | 2.96 [1.87 to 3.58] | 3.02 [1.74 to 3.98]
Statistical Analysis 1: Comparison: Pemetrexed + Enzastaurin vs Pemetrexed + Placebo; Test type: Superiority or Other; p = 0.544, Log Rank — P-value was stratified by Eastern Cooperative Oncology Group (ECOG) performance status and time since last chemotherapy; Hazard Ratio (HR) = 1.13, 95% CI [0.77 to 1.65]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of randomization to the date of death from any cause. For participants who were alive at the time of the data inclusion cutoff, OS was censored at the date the participant was last known to be alive.
Time Frame: Baseline to date of death from any cause up to 12.32 months
Population: All randomized participants. Fifty three (53) participants in Pemetrexed + Enzastaurin group and forty five (45) participants in Pemetrexed + Placebo group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 80 | 80
months | 9.63 [8.18 to NA] — Upper limit of 95% confidence interval was not estimable due to high censoring rate. | 7.39 [6.41 to NA] — Upper limit of 95% confidence interval was not estimable due to high censoring rate.
Statistical Analysis 1: Comparison: Pemetrexed + Enzastaurin vs Pemetrexed + Placebo; Test type: Superiority or Other; p = 0.171, Log Rank — P-value was stratified by Eastern Cooperative Oncology Group (ECOG) performance status and time since last chemotherapy; Hazard Ratio (HR) = 0.70, 95% CI [0.42 to 1.17]

3. Secondary Outcome: Time-to-Worsening (TW) in Lung Cancer Symptom Scale (LCSS) - Health Related Quality of Life (HRQoL) Subscale
Description: LCSS is a participant rated lung cancer instrument which consisted of 6 disease related symptoms (appetite, cough, fatigue, dyspnea, hemoptysis, and pain) and 3 quality of life (QoL) items (activity status, symptomatic distress, and overall QoL). TW in LCSS-HRQoL was measured from the date of enrollment to the first date of a 15 millimeters (mm) worsening in the 9th LCSS item on QoL. LCSS-HRQoL was measured on the 100-mm visual analogue scale (VAS) with the scores ranging from 0 (best response and very high HRQoL) to 100-mm (worse response and very low HRQoL). TW-HRQoL was censored at the date of the participant's last LCSS assessment for participant without a 15-mm increase on the 100-mm VAS.
Time Frame: Baseline to disease worsening up to 10.58 months
Population: Randomized participants who had at least 1 baseline and 1 postbaseline LCSS assessment for HRQoL. Thirty (30) participants in Pemetrexed + Enzastaurin group and forty (40) participants in Pemetrexed + Placebo group were censored for the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 63 | 61
months | 3.06 [2.37 to 4.63] | 8.08 [3.81 to NA] — Upper limit of 95% confidence interval was not estimable due to high censoring rate.
Statistical Analysis 1: Comparison: Pemetrexed + Enzastaurin vs Pemetrexed + Placebo; Test type: Superiority or Other; p = 0.010, Regression, Cox; Hazard Ratio (HR) = 2.11, 95% CI [1.19 to 3.75]

4. Secondary Outcome: Duration of Disease Control (DDC)
Description: DDC was defined as the time from randomization to the first documented observation of disease progression or death from any cause and was limited to the participants with a best tumor response of complete response (CR), partial response (PR), or stable disease (SD). Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive disease (PD) was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. SD was defined as small changes that did not meet the above criteria. DDC was censored at the date of the last objective progression-free disease assessment for participants who did not experience PD or death.
Time Frame: Baseline to measured progressive disease up to 9.92 months
Population: Randomized participants who received at least 1 dose of study drug and had a best tumor response of CR, PR, or SD. Fourteen (14) participants in Pemetrexed + Enzastaurin group and seventeen (17) participants in Pemetrexed + Placebo group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 38 | 38
months | 5.32 [3.58 to 7.13] | 6.31 [4.40 to 6.93]
Statistical Analysis 1: Comparison: Pemetrexed + Enzastaurin vs Pemetrexed + Placebo; Test type: Superiority or Other; p = 0.194, Log Rank — P-value was stratified by Eastern Cooperative Oncology Group (ECOG) performance status score and time since last chemotherapy; Hazard Ratio (HR) = 1.50, 95% CI [0.81 to 2.77]

5. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Tumor Response Rate)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Participants with a best response of complete response (CR) or partial response (PR) were considered to have had a tumor response. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Percentage of participants was calculated as the total number of participants affected divided by the number of participants analyzed then multiplied by 100.
Time Frame: Baseline to measured progressive disease up to 9.92 months
Population: Randomized participants who received at least 1 dose of study drug and had responses evaluated for CR or PR.
Measure: Number; unit: percentage of participants
Groups:
- Pemetrexed + Enzastaurin: Enzastaurin 1125 milligrams (mg) loading dose [total 9 tablets; three (125-mg) tablets administered orally 3 times a day] on Day 1 followed by total dose of 500 mg enzastaurin [two (125-mg) tablets administered orally 2 times a day] on Days 2 to 28, and pemetrexed 500 milligrams per square meter (mg/m^2) intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by total dose of 500 mg enzastaurin [two (125-mg) tablets administered orally 2 times a day] on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Pemetrexed + Placebo: Placebo loading dose (total 9 tablets; three tablets administered orally 3 times a day) on Day 1 followed by four placebo tablets (two tablets 2 times a day) on Days 2 to 28, and pemetrexed 500 mg/m^2 intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by four placebo tablets (two tablets 2 times a day) on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
  .
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 77 | 78
percentage of participants | 3.9 | 2.6
Statistical Analysis 1: Comparison: Pemetrexed + Enzastaurin vs Pemetrexed + Placebo; Test type: Superiority or Other; p = 0.681, Fisher Exact

6. Secondary Outcome: Tumor Biomarkers
Description: Protein expression was measured using an Immunohistochemistry (IHC) assay from the tumor tissue samples. IHC histo-scores (H-scores) were determined separately for each of the 3 biomarkers: folate receptor alpha (FR alpha) in cytoplasm and apical membrane, thymidylate synthase (TS) in cytoplasm and nucleus, and thyroid transcription factor-1 (TTF1) in the nucleus. Tumor tissue samples were to be scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system for cytoplasmic and nuclear staining. IHC H-score was calculated using the formula: 1 * (percentage of cells stained 1+) + 2 * (percentage of cells stained 2+) + 3 * (percentage of cells stained 3+), giving a minimum score of 0 to a maximum score of 300. The maximum score indicates the strongest expression.
Time Frame: Tumor samples collected at baseline
Population: Randomized participants who had at least 1 biomarker expression value measured at baseline.
Measure: Mean (Standard Deviation); unit: H-scores
Groups:
- Total (Pemetrexed + Enzastaurin and Pemetrexed + Placebo): Enzastaurin (1125 mg loading dose of 9 tablets) or placebo (loading dose of 9 tablets) administered on Day 1 followed total dose of 500 mg enzastaurin (two 125-mg tablets administered orally 2 times a day) or four placebo tablets (2 tablets 2 times a day) on Days 2 to 28, and pemetrexed 500 mg/m^2 intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by total dose of 500 mg enzastaurin [two 125-mg tablets administered orally 2 times a day] or four placebo tablets (2 tablets 2 times a day) on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo | Total (Pemetrexed + Enzastaurin and Pemetrexed + Placebo)
Number analyzed (Participants) | 26 | 20 | 46
H-scores
  FR Alpha in Cytoplasm: number analyzed (Participants) | 25 | 20 | 45
  FR Alpha in Cytoplasm | 55.96 (65.99) | 24.50 (51.04) | 41.98 (61.24)
  FR Alpha in Apical Membrane: number analyzed (Participants) | 25 | 20 | 45
  FR Alpha in Apical Membrane | 9.96 (24.70) | 18.25 (48.62) | 13.64 (37.03)
  TS in Cytoplasm | 16.38 (25.29) | 22.30 (34.83) | 18.96 (29.60)
  TS in Nucleus | 5.92 (12.55) | 8.00 (18.84) | 6.83 (15.44)
  TTF-1 in Nucleus | 47.88 (71.18) | 32.35 (72.58) | 41.13 (71.41)

7. Other Pre Specified Outcome: Number of Participants Who Died During the Study Treatment
Description: Reported are the deaths due to study disease and adverse events (AEs) that occurred while on study treatment.
Time Frame: Baseline through study completion [up to 16 Cycles (21-day cycles, except Cycle 1 [28 days])]
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 79 | 80
Participants
  Study Disease | 2 | 3
  AEs | 1 | 3

8. Other Pre Specified Outcome: Number of Participants Who Died During the 30 Days After Treatment Discontinuation
Description: Reported are the deaths due to study disease and adverse events (AEs) that occurred during the 30 days after treatment discontinuation.
Time Frame: End of study treatment [16 Cycles (21-day cycles, except Cycle 1 [28 days])] through 30 days after treatment discontinuation
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pemetrexed + Placebo: Placebo loading dose [total 9 tablets (3 tablets administered orally 3 times a day)] on Day 1 followed by 4 placebo tablets (2 tablets 2 times a day) on Days 2 to 28, and pemetrexed 500 mg/m^2 intravenous injection on Day 8 in Cycle 1 (28-day cycle).
  Pemetrexed 500 mg/m^2 intravenous injection on Day 1 followed by 4 placebo tablets (2 tablets 2 times a day) on Days 1 to 21 in Cycle 2 and subsequent cycles (21-day cycle).
  Treatment was continued until evidence of disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
  .
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Number analyzed (Participants) | 79 | 80
Participants
  Study Disease | 5 | 10
  AEs | 2 | 0

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease (PD) were not considered to be serious adverse events (SAEs) unless the investigator deemed it related to the use of the study drug.
Arm/Group | Pemetrexed + Enzastaurin | Pemetrexed + Placebo
Serious Adverse Events (participants affected / at risk) | 33/79 | 30/80
Other Adverse Events (participants affected / at risk) | 73/79 | 75/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Enzastaurin (N=79) | Pemetrexed + Placebo (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 5 (5) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 1 (1)
Listeriosis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 4 (6)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Enzastaurin (N=79) | Pemetrexed + Placebo (N=80)
Anaemia (Blood and lymphatic system disorders) | 23 (26) | 15 (22)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 3 (8)
Lymphopenia (Blood and lymphatic system disorders) | 5 (9) | 5 (7)
Neutropenia (Blood and lymphatic system disorders) | 15 (16) | 6 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (18) | 5 (14)
Vertigo (Ear and labyrinth disorders) | 5 (7) | 4 (4)
Lacrimation increased (Eye disorders) | 7 (7) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 8 (11)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 4 (5)
Constipation (Gastrointestinal disorders) | 19 (20) | 16 (19)
Diarrhoea (Gastrointestinal disorders) | 17 (25) | 11 (13)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (6)
Nausea (Gastrointestinal disorders) | 38 (52) | 20 (29)
Vomiting (Gastrointestinal disorders) | 19 (25) | 14 (18)
Asthenia (General disorders) | 19 (22) | 17 (26)
Chest pain (General disorders) | 9 (9) | 11 (11)
Fatigue (General disorders) | 23 (29) | 24 (27)
General physical health deterioration (General disorders) | 2 (2) | 5 (5)
Mucosal inflammation (General disorders) | 8 (13) | 5 (5)
Oedema (General disorders) | 4 (5) | 3 (3)
Oedema peripheral (General disorders) | 11 (13) | 8 (9)
Pyrexia (General disorders) | 16 (28) | 14 (18)
Candidiasis (Infections and infestations) | 7 (7) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 5 (8)
Platelet count decreased (Investigations) | 4 (4) | 1 (1)
Weight decreased (Investigations) | 9 (9) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 28 (37) | 15 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Dizziness (Nervous system disorders) | 10 (13) | 5 (5)
Headache (Nervous system disorders) | 7 (8) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 5 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 7 (7) | 8 (13)
Chromaturia (Renal and urinary disorders) | 8 (8) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 16 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 15 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 13 (16) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days